CLINICAL TRIAL: NCT00911131
Title: A New Technique to Enhance Detection of Small Esophageal Varices by PillCam ESO Capsule Endoscopy
Brief Title: Enhancing Detection of Small Esophageal Varices by PillCam ESO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Kia Saeian, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRO 8503
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Esophageal Varices
Keywords: Small grade esophageal varices; capsule endoscopy; PillCam ESO; abdominal binder
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Screening esophagoduodenoscopy (EGD) (Active Comparator): EGD will be performed utilizing conscious sedation. During EGD, the endoscopist will capture pictures of the esophageal body, Z-line, lower esophagus and proximal gastric folds. Grading of esophageal varices will be performed by all investigators using the Italian Liver cirrhosis project.
  Patients who are found to have small grade varices and meet the inclusion and exclusion criteria will be enrolled in the study.
  Interventions: Procedure: EGD
- Capsule Endoscopy (Active Comparator): The capsule endoscope will be swallowed by the participant with 100cc of water and simethicone in the supine position. Recording is done for 2 minute in this position and then the head will be elevated to 30 degrees for 2 minutes and then 60 degrees for 1 minute. After 1 minute, the patient will sip10cc of water and after 15 seconds, they will sit upright and sip water again. They can then walk and resume normal activity for 15 minutes. The videos will be reviewed and graded by a gastroenterologist experienced with capsule endoscopy and will be blinded to the patient's clinical and procedural history as well as the most recent EGD. The varices will be graded using the Given Imaging software that grades varices as no varices (C0), small varices or < 25% of esophageal circumference (C1), and large varices or > 25% of esophageal circumference (C2).
  Interventions: Device: Capsule endoscopy (PillCam ESO)
- Capsule Endoscopy with abdominal binder (Active Comparator): Before swallowing the capsule endoscope, an inflatable girdle is wrapped around the waist above the umbilicus and held in place by a an abdominal binder. The pressure is increased by 10mmHg for 10 minutes. The PillCam ESO is placed in the mouth and the patient is asked to swallow it with 100cc of water with simethicone in the supine position. Recording is done for 2 minute in this position and then the head is elevated to 30 degrees for 2 minutes and then 60 degrees for 1 minute. After 1 minute, the patient sips 10cc of water and after 15 seconds, they sit upright and sip water again. They can then walk and resume normal activity for 15 minutes.
  Interventions: Device: Capsule endoscopy (PillCam ESO) with abdominal binder

INTERVENTIONS:
Device: Capsule endoscopy (PillCam ESO) — The capsule endoscope is placed in the mouth and the patient is asked to swallow it with 100cc of water with simethicone in the supine position. Recording is done for 2 minute in this position and then the head is elevated to 30 degrees for 2 minutes and then 60 degrees for 1 minute. After 1 minute, the patient sips 10cc of water and after 15 seconds, they sit upright and sip water again. They can then walk and resume normal activity for 15 minutes.
  Other Names: PillCam ESO
  Arms: Capsule Endoscopy
Procedure: EGD — Patients will undergo conventional EGD under conscious sedation for routine screening of esophageal varices.
  Other Names: Esophagoduodenoscopy
  Arms: Screening esophagoduodenoscopy (EGD)
Device: Capsule endoscopy (PillCam ESO) with abdominal binder — An abdominal binder with and inflatable girdle is wrapped around the stomach prior to swallowing the capsule endoscope. The girdle is inflated to 10mmHg for 10 minutes. The capsule is swallowed by the patient and the routine method for the procedure is performed.
  Other Names: PillCam ESO
  Arms: Capsule Endoscopy with abdominal binder

SUMMARY:
Increasing intra-abdominal pressure (IAP) with an abdominal binder will increase pressure within smaller esophageal varices which will therefore enhance the ability of capsule endoscopy to detect these varices better.

Therefore, the aims of the investigators' study are as follows:

1. To determine if using an abdominal binder to increase IAP can increase the detection rate of small esophageal varices when using capsule endoscopy.
2. To determine if using an abdominal binder to increase IAP during capsule endoscopy has a comparable detection rate of small esophageal varices to conventional endoscopy.

DETAILED DESCRIPTION:
Esophageal variceal bleeding is a common and life-threatening complication of portal hypertension in patients with cirrhosis of liver. It is associated with a mortality rate of up to 50% in these patients. Prophylactic treatments to prevent variceal bleeding, therefore, assume paramount clinical significance. Currently, primary prophylactic treatments using pharmacologic agents with non-selective beta blockers as well as endoscopic variceal ligation (EVL) are effectively employed in preventing variceal bleeding. The American Association for the Study of Liver Disease (AASLD) guidelines recommend that patients with Child's stage A cirrhosis and portal hypertension with platelet count less than 140,000/mmq or portal vein diameter > 13mm and those patients classified as Child's B and C cirrhosis should undergo screening endoscopy for esophageal varices. Patients with cirrhosis and no esophageal varices detected during screening should undergo endoscopy ever three years. Patients with small esophageal varices are recommended to be screened endoscopically every 1 to 2 years.

Currently, esophagogastroduodenoscopy (EGD) under conscious sedation is the gold standard for variceal screening. However, EGD has certain limitations especially when used in patients with cirrhosis of the liver. Prolonged conscious sedation may have an adverse effect on encephalopathy. EGD also may not be cost effective for screening esophageal varices.

The use of PillCam ESO capsule endoscopy to detect esophageal varices has become an attractive alternative to conventional endoscopy especially in patients unwilling to undergo EGD. Identifying patients with small varices, which have the potential for progression to large varices and bleeding, is an important clinical issue to address.

ELIGIBILITY:
Inclusion Criteria:

* patients identified with grade I and grade II esophageal varices by conventional endoscopy who are returning for screening or surveillance
* patients who have had endoscopic banding of varices in the past
* patients aged 18 years or older
* patients able to give consent
* patients eligible and willing to undergo upper endoscopy and PillCam ESO capsule endoscopy

Exclusion Criteria:

* dysphagia
* Zenker's diverticulum
* pregnancy
* esophageal stricture
* gastric or intestinal obstruction
* multiple abdominal surgeries
* cardiac pacemakers
* implanted electronic medical devices
* cognitive impairment
* also, patients found to have bleeding, requiring banding, or other complications on screening EGD the day of the trial will not proceed to capsule endoscopy
* urine pregnancy test will be conducted prior to participation; this is part of the standard procedure for women of child-bearing age undergoing upper endoscopy in the GI lab
* all patients being evaluated for the current study will be evaluated for the presence or absence of overt portosystemic encephalopathy:

  * Those found to have overt portosystemic encephalopathy will then be graded based on the standard scale of grade 1 through 4 portosystemic encephalopathy. Assessment of whether patients with liver disease and hepatocellular carcinoma possess decisional capacity is essentially the same as for other subjects with the exception that due diligence must be used to address whether there is any evidence of active ongoing overt portosystemic encephalopathy. From the available data and current standards of care, patients with stage 1 overt hepatic encephalopathy are decisional but may have minimal impairment in their cognitive skills particularly in the domains of attention and sleep. Decisional capacity in patients with grades 2-4 overt portosystemic encephalopathy is impaired and will lead to them bring excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Detection rate of esophageal varices using different screening modalities. | 30 days

SECONDARY OUTCOMES:
Patient tolerability of each screening modality. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kia Saeian, MD, Study Director — Medical College of Wisconsin; Mukund Venu, MD, Principal Investigator — Medical College of Wisconsin

REFERENCES:
- [Background] D'Amico G, Pagliaro L, Bosch J. Pharmacological treatment of portal hypertension: an evidence-based approach. Semin Liver Dis. 1999;19(4):475-505. doi: 10.1055/s-2007-1007133. PMID 10643630
- [Background] Christensen E, Fauerholdt L, Schlichting P, Juhl E, Poulsen H, Tygstrup N. Aspects of the natural history of gastrointestinal bleeding in cirrhosis and the effect of prednisone. Gastroenterology. 1981 Nov;81(5):944-52. PMID 7026343
- [Background] Grace ND, Groszmann RJ, Garcia-Tsao G, Burroughs AK, Pagliaro L, Makuch RW, Bosch J, Stiegmann GV, Henderson JM, de Franchis R, Wagner JL, Conn HO, Rodes J. Portal hypertension and variceal bleeding: an AASLD single topic symposium. Hepatology. 1998 Sep;28(3):868-80. doi: 10.1002/hep.510280339. No abstract available. PMID 9731585
- [Background] de Franchis R. Updating consensus in portal hypertension: report of the Baveno III Consensus Workshop on definitions, methodology and therapeutic strategies in portal hypertension. J Hepatol. 2000 Nov;33(5):846-52. doi: 10.1016/s0168-8278(00)80320-7. No abstract available. PMID 11097497
- [Background] Assy N, Rosser BG, Grahame GR, Minuk GY. Risk of sedation for upper GI endoscopy exacerbating subclinical hepatic encephalopathy in patients with cirrhosis. Gastrointest Endosc. 1999 Jun;49(6):690-4. doi: 10.1016/s0016-5107(99)70283-x. PMID 10343210
- [Background] Saeian K, Staff D, Knox J, Binion D, Townsend W, Dua K, Shaker R. Unsedated transnasal endoscopy: a new technique for accurately detecting and grading esophageal varices in cirrhotic patients. Am J Gastroenterol. 2002 Sep;97(9):2246-9. doi: 10.1111/j.1572-0241.2002.05906.x. PMID 12358240
- [Background] Eisen GM, Eliakim R, Zaman A, Schwartz J, Faigel D, Rondonotti E, Villa F, Weizman E, Yassin K, deFranchis R. The accuracy of PillCam ESO capsule endoscopy versus conventional upper endoscopy for the diagnosis of esophageal varices: a prospective three-center pilot study. Endoscopy. 2006 Jan;38(1):31-5. doi: 10.1055/s-2005-921189. PMID 16429352
- [Background] Lapalus MG, Dumortier J, Fumex F, Roman S, Lot M, Prost B, Mion F, Ponchon T. Esophageal capsule endoscopy versus esophagogastroduodenoscopy for evaluating portal hypertension: a prospective comparative study of performance and tolerance. Endoscopy. 2006 Jan;38(1):36-41. doi: 10.1055/s-2006-924975. PMID 16429353
- [Background] Pena LR, Cox T, Koch AG, Bosch A. Study comparing oesophageal capsule endoscopy versus EGD in the detection of varices. Dig Liver Dis. 2008 Mar;40(3):216-23. doi: 10.1016/j.dld.2007.10.022. Epub 2007 Dec 21. PMID 18082473
- [Background] de Franchis R, Eisen GM, Laine L, Fernandez-Urien I, Herrerias JM, Brown RD, Fisher L, Vargas HE, Vargo J, Thompson J, Eliakim R. Esophageal capsule endoscopy for screening and surveillance of esophageal varices in patients with portal hypertension. Hepatology. 2008 May;47(5):1595-603. doi: 10.1002/hep.22227. PMID 18435461
- [Background] Merli M, Nicolini G, Angeloni S, Rinaldi V, De Santis A, Merkel C, Attili AF, Riggio O. Incidence and natural history of small esophageal varices in cirrhotic patients. J Hepatol. 2003 Mar;38(3):266-72. doi: 10.1016/s0168-8278(02)00420-8. PMID 12586291
- [Background] Luca A, Cirera I, Garcia-Pagan JC, Feu F, Pizcueta P, Bosch J, Rodes J. Hemodynamic effects of acute changes in intra-abdominal pressure in patients with cirrhosis. Gastroenterology. 1993 Jan;104(1):222-7. doi: 10.1016/0016-5085(93)90855-7. PMID 8419245
- [Background] Escorsell A, Gines A, Llach J, Garcia-Pagan JC, Bordas JM, Bosch J, Rodes J. Increasing intra-abdominal pressure increases pressure, volume, and wall tension in esophageal varices. Hepatology. 2002 Oct;36(4 Pt 1):936-40. doi: 10.1053/jhep.2002.35817. PMID 12297841